CLINICAL TRIAL: NCT03559127
Title: Pain Reduction After One-visit Root Canal Treatment Using Two Cold Irrigating Protocols in Teeth With Vital Pulps.
Brief Title: Pain Reduction Using Two Cold Irrigating Protocols in Teeth With Vital Pulps.
Acronym: EP18
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Jorge Paredes Vieyra, DDS, MsC, PhD, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Pain after RCT 2018
Record Dates: First submitted 2018-05-10; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Post Operative Pain
Keywords: post-endodontic pain; pain; criotherapy; cold irrigation
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Random Selection of different temperature of irrigating solution groups. Of the sample of 240 teeth, 80 were randomly assigned to the one of the 3 irrigating protocols. Treatment was performed by 3 experienced endodontists; each prepared and irrigated 80 teeth.
Who Masked: Participant, Investigator
Masking Description: Certified endodontist (3) trained in the procedures, devices, and irrigating systems investigated took part in the research. All experts tracked a pre-established procedure for Reciproc instrument systems and cryotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A. Cold Protocol with 6 oC (Experimental): Use of 20 mL cold (6 oC) sterile saline solution.
  After the clinical procedure cryotherapy was applied. 5 mL cold (6 oC) 17% EDTA followed with 20 mL cold (6 oC) sterile saline solution dispensed to the WL using a cold (6 oC) metallic micro-cannula included in the Endo Vac System for five minutes.
  Interventions: Procedure: For the Group A. Applied Cryotherapy at 6 oC
- Group B. Cold Protocol with 2.5 oC (Experimental): Use of 20 mL cold (2.5 oC) sterile saline solution
  After the procedure cryotherapy was applied. 5 mL cold (2.5 oC) 17% EDTA followed with 20 mL cold (2.5 oC) sterile saline solution dispensed to the WL using a cold (2.5 oC) metallic micro-cannula included in the Endo Vac System for five minutes.
  Interventions: Procedure: For the Group B. Applied Cryotherapy at 2.5 oC
- CG. Room temperature Protocol (Experimental): Use of 20 mL (at room temperature) sterile saline solution
  The group will receive irrigant at room temperature. 5mL of 17% EDTA and 20 mL of sterile saline usingmetallic micro-cannula included in the Endo Vac System for five minutes.
  Interventions: Procedure: Control Group (CG). Applied irrigant at room temperature

INTERVENTIONS:
Procedure: For the Group A. Applied Cryotherapy at 6 oC — Patients assigned to this group receive a final irrigation with 5 mL cold (6 oC) 17% EDTA followed with 20 mL cold (6 oC) sterile saline solution dispensed to the WL using a cold (6 oC) metallic micro-cannula included in the Endo Vac System (Kerr Endo) for 5 minutes.
  Other Names: Cold irrigant used after root canal treatment
  Arms: Group A. Cold Protocol with 6 oC
Procedure: For the Group B. Applied Cryotherapy at 2.5 oC — Patients assigned to this group receive a final irrigation with 5 mL cold (2.5 oC) 17% EDTA followed with 20 mL cold (2.5 oC) sterile saline solution dispensed to the WL using a cold (2.5 oC) metallic micro-cannula included in the Endo Vac System for five minutes.
  Other Names: Cold irrigant used after RCT
  Arms: Group B. Cold Protocol with 2.5 oC
Procedure: Control Group (CG). Applied irrigant at room temperature — Patients assigned to this control group were treated identically to the experimental groups, except that receive a final flush with 5 mL (room temperature) 17% EDTA followed with twenty mL (room temperature) sterile saline solution delivered to the WL using a metallic micro-cannula included in the Endo Vac System for five minutes.
  Other Names: Use of Saline solution at room temperature
  Arms: CG. Room temperature Protocol

SUMMARY:
The goal of this clinical research was to relate the incidence of post-endodontic pain after one-visit root canal treatment using two cold protocols of irrigation. Methodology: All 240 patients had upper or lower molar, premolar or anterior teeth selected for conventional root canal treatment for prosthetic reasons detected with only vital pulps (symptomatic or asymptomatic condition). Of the sample of 240 teeth, were selected to different manner to irrigate. Reciproc instruments were used with a micro motor (VDW, Munich Germany). Final irrigation with cold (6oC, 2.5 oC and room temperature 17% EDTA and saline solution served as a lubricants.

DETAILED DESCRIPTION:
RCT was done in one-visit. Topical anesthetic (Anestesia Topica, Astra Mexico) was applied before infiltration. Patients received 2 carpules of articaine 2% with epinephrine 1:200,000 (Septodont, Saint-Maur des-Fosses, France). In circumstances in which additional anesthesia was required, intra-ligamental anesthesia (2 mL articaine 2%) was administered. For the upper teeth, the solution was injected by slow and gradual local infiltration. For the lower teeth, 1 of the carpules was used for an inferior alveolar nerve block and the other 1 for a gentle labial infiltration near the tooth to be treated.

Rubber dam was placed and the tooth was clean with 5.25% NaOCl. Preparation of the access cavity was achieved using sterile # 331 bur (Dentsply Int, York, PA), with high-speed and refrigeration. 5.25% NaOCl was employed to disinfect the coronal access. The canals were cautiously probed with #10 K-type file (Flex-R files, Moyco/Union Broach, York PA, USA).

17% EDTA (Roth International, Chicago, IL) irrigant was administered at the entrance of the canals. Working length was established with a #15 k-file and the Root ZX electronic apex locator (J Morita, Irvine CA, USA), and confirmed radiographically (Schick Technologies, NY, USA). Cervical and middle thirds of the canal was flared with a K3XF 25/10 rotary instrument (Kerr Endo, Orange County, CA) at 500 rpm. The root canal was flushed with 3 mL 5.25% sodium hypochlorite (NaOCl). A glide path to the WL was then established.

Preparations of the canals were completed with an electric motor (VDW Silver Motor, VDW, Munich Germany). Torque and rotation were predetermined for each reciproc instrument, and were used in continuous reciprocating mode.

Dentinal remains were removed from the instrument with a sterile gauze, immediately to the instrument change after two-three pull in-and-pull out (pecking) movements (Reciproc) following the manufacturers' recommendations.

Each root canal was flushed with 2.5mL 2.6% NaOCl. Irrigation was achieved using a 24-gauge needle (Max-I-Probe; Tulsa Dental, York, PA) and a 31-G NaviTip needle (Ultradent Products Inc, South Jordan, UT) when getting the WL after each instrument insertion. A size #10 K file was used to maintain WL after each Reciproc instrument. The established WL was checked repeatedly throughout the clinical procedures.

After instrumentation, the root canals were flushed with 1 mL 2.6% NaOCl, activated ultrasonically; It was achieved by means of an Irrisafe ultrasonic 20.00 tip (Satelec, Merignac, France) at 50% power of the Mini-Endo ultrasonic device (Kerr Endo) with the tip placed three mm from the WL for thirty seconds per root canal.

Irrigating Protocols Group A. The R25 (size 25/ .08) instrument was used in thin and curved canals, and R40 files (40/ .06) were used in broad root canals. Three in/out pecking cycles were employed with a fullness of not more than 3 mm until reaching the established WL. Patients assigned to this group receive a final irrigation with 5 mL cold (6 oC) 17% EDTA followed with 20 mL cold (6 oC) sterile saline solution dispensed to the WL using a cold (6 oC) metallic micro-cannula included in the Endo Vac System (Kerr Endo) for 5 minutes.

Group B. Canals were prepared as in group A, Patients assigned to this group receive a final irrigation with 5 mL cold (2.5 oC) 17% EDTA followed with 20 mL cold (2.5 oC) sterile saline solution dispensed to the WL using a cold (2.5 oC) metallic micro-cannula included in the Endo Vac System for five minutes.

Control Group (CG). The R25 (size 25/ .08) instrument was used in thin and curved root canals, and R40 files (40/ .06) were used in wide root canals. Three in-and-out cycles were applied with a distance of not more than three mm until getting the established WL. Reciproc instruments were employed in one tooth only (single use). Patients assigned to this control group were treated identically to the experimental groups, except that receive a final flush with 5 mL (room temperature) 17% EDTA followed with twenty mL (room temperature) sterile saline solution delivered to the WL using a metallic micro-cannula included in the Endo Vac System for five minutes.

Each experimental and control group were flushed with the irrigant described above. Care was taken to confirm that the metallic cannula would aspirate properly by noticing the system's translucent evacuation duct. In case there was some obstacle, the metallic device was rapidly replaced.

Recapitulation of working length was performed again by using an apex locator as described before using #35 and #40 files.

The root canals were desiccated with disinfected paper cones and filled at the same visit. Gutta-percha points (Dentsply Maillefer) were laterally condensed with #25 nickel-titanium spreaders (Dentsply Maillefer) and AH-plus as the sealer (Dentsply Maillefer). The access cavities were etched and fixed with Fuji IX (GC Corp, Tokyo, Japan).

After these irrigation regimens, the patients were warned of the possible occurrence of pain for hours following RCT and received an evaluation form (VAS questionnaire) to be completed and give it back 72 hours after. In it, they confirmed the presence/absence of pain. The pain level was measured using a validated pain scale known as the VAS (Hawker et al. 2011). The VAS scale is a continuous measure comprised of a horizontal line, which is 10 cm in length. For pain intensity, the VAS is anchored by ''no pain'' (score of 0) and ''pain as bad as it could be'' (score of 10). The cut points on the pain VAS are no pain (0-0.5 cm), mild pain (0.6-4.0 cm), moderate pain (0.45-7.4 cm), and severe pain (7.5-10 cm) (Jensen et al. 2003). The pain VAS was completed by the patients. The patients were asked to put a mark perpendicular to the pain VAS line at the point that indicated their pain severity during the 3 days after the endodontic treatment.

234 of the two hundred and forty examinations were properly returned. 77 belonged to the group A, 78 to group B and 79 to the Control group. The missing 6 questionnaires were returned one day later and were incorporated in the examination.

The outcomes for the groups A, B and CG related to existence (yes/no), kind (mild, moderate, severe), and period (days) of pain were evaluated, and related to the following diagnostic factors: vital teeth, presence or absence of pre-operative pain, group of teeth, or ubication, age and sex, presence of occlusal contacts.

ELIGIBILITY:
Inclusion Criteria:

- absence of radiographic sign of apical pathosis and a diagnosis of irreversible pulpitis (IP) and vital pulp established by affirmative response to hot and cold examinations.

* Thermal pulp examination was achieved by the corresponding author, and radiographic analysis was established by 3 certified endodontists.
* Clinical requirements were established on the next conditions: 1) The purposes and necessities of the research were spontaneously accepted. 2) Clinical Management was pointed to patients in physical and mental well- being. 3) All teeth had vital pulps and absence of apical periodontitis. 4) Positive thermal stimulation with EndoIce (Hygenic Corp, Akron, OH). 5) Teeth with enough coronal structure for rubber dam isolation. 6) No root canal therapy done before the research. 7) No painkillers or antibiotics used 7 days' prior the clinical events started.

Exclusion Criteria:

* the necessity for retreatment

  * pregnancy
  * impossibility to obtain patient's approval
  * patients who didn't complete inclusion necessities for the research
  * a history of medication for chronic pain or those compromising the immune response
  * patients younger than 18 years and the existence of mishaps or difficulties during RCT (calcified canals, impracticality of achieving Apical patency).

Root fractures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the post-endodontic pain after one-visit after the root canal treatment with reciprocating NiTi system. | 24 hours to 72 hours
  Pain was evaluated after 24, 48 and 72 hrs after instrumentation with reciproc NiTi instruments, the 80 canals were flushed with cold irrigants (6 and 2.5 oC). According to the VAS table provided to the participants

SECONDARY OUTCOMES:
Evaluate the Use of intracanal cryotherapy on post-endodontic pain after single-visit RC. | 24 hours to 72 hours
  Pain reduction was evaluated after a final irrigation with cold 5cc of (2.5 oC- 6 oC) 17% EDTA gently delivered to the WL using a cold (2.5- 6 oC) sterile metallic micro cannula. According to the VAS table provided to the participants

CONTACTS AND LOCATIONS:
Locations (3):
- Mexico (3):
  - Jorge Paredes Vieyra, Tijuana, Baja Califronia
  - Jorge Paredes Vieyra, Tijuana, Estado de Baja California
  - Jose Clemente, Tijuana, Estado de Baja California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729